CLINICAL TRIAL: NCT07207538
Title: Impact of Physical Exercise on Telomere Length and Other Markers of Premature Ageing in First-episode Psychosis.
Brief Title: Physical Exercise in Patients With First Psychotic Episode
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Juan Luis Sanchez Gonzalez, Principal investigator. Juan Luis Sánchez González, University of Salamanca
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ExerciseFirstPsychoticEpisode
Record Dates: First submitted 2025-09-23; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Telomere Length; Exercise; First Episode Psychosis (FEP)
Keywords: Exercise; Telomere length; Aging
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The persons in charge of the evaluation of the participants will be unaware of the assignment of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention group (Experimental): n additional strength training programme will be carried out for 12 weeks with 2 sessions per week. The sessions will last approximately 50 minutes and will be divided into 3 distinct parts: The first part will consist of a warm-up with a part of aerobic exercise that will last approximately 15 minutes. This will be followed by the main part of strength training with a circuit of 6 exercises (3 series x 12 repetitions) which will last approximately 25 minutes. Finally, there will be a cool down phase with breathing exercises to allow people to recover.
  Interventions: Other: Other: Strength physical exercise programme
- Sham Comparator: Control group (Sham Comparator): Subjects in the control group will continue with their normal life and carry out all the activities they have been doing previously.
  Interventions: Other: Other: Normal life

INTERVENTIONS:
Other: Other: Strength physical exercise programme — 12 multi-joint strength exercises will be developed. Participants will be taught the rating scale of perceived exertion (RPE) based on the number of repetitions in reserve (RIR). Participants will be asked that during the performance of each of the exercises they must perceive an effort between 7-8 within the overall score of the scale (0-10; 0 = no effort at all and 10 = cannot perform one more repetition, i.e. maximal effort). When subjects perform the 12 repetitions with lower perceived exertion than the set effort in two consecutive sessions with full range of motion the training load will be increased by about 2-10% following the American College of Sports Medicine guidelines and reassessed using the RIR-based RPE. Patients in the usual treatment group will continue to participate in their existing rehabilitation programmes, but will not be included in the strength training programme.
  Arms: Experimental: Intervention group
Other: Other: Normal life — Description: Normal life and carry out all the activities they have been doing previously.
  Arms: Sham Comparator: Control group

SUMMARY:
Justification: Patients with first-episode psychosis are at increased risk of premature ageing and early mortality, associated with telomere shortening and increased inflammatory markers. Physical exercise has shown protective effects in the general population, but there are no intervention studies in this population.

Objective: To evaluate the effect of a strength training programme on telomere length and other markers of cellular ageing in people with a first episode of psychosis.

Material and methods: Quasi-experimental study with patients aged 18-35 years included in the PRINT programme (Salamanca). Standard treatment will be compared with standard treatment plus a 12-week strength training programme. Telomere length (qPCR), inflammatory and senescence markers (proteomics), body composition, frailty and quality of life will be analysed.

Applicability: The results could support the inclusion of physical exercise programmes as a complementary intervention in early psychosis care, promoting overall health, quality of life and reducing the gap in life expectancy compared to the general population.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* Having experienced a first psychotic episode in the last 3 years

Exclusion Criteria:

* are unable to read and understand the patient information sheet and sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Telomere Length | Baseline and immediately after the intervention
  Telomere length will be measured before and after the procedure in kilobases.

SECONDARY OUTCOMES:
Fragility | Baseline and immediately after the intervention
  Fragility will be measured using the Short Physical Performance Battery scale (SPPB). SPPB scores range from zero to 12 possible points. SPPB score of 3-9 points in persons with possible sarcopenia but no mobility disability indicates frailty; SPPB score of 10 or greater for persons with no sarcopenia and no mobility disability indicates robustness. Persons with a score of 2 or lower who have sarcopenia, potential cachexia, and mobility disability are determined to be disabled.
Quality of life | Baseline and immediately after the intervention
  Quality of life will be assessed using the EuroQuality of Life (EQ-5D-5L scale). This scale is numbered from 0 to 100. • 100 means the best health you can imagine. 0 means the worst health you can imagine.
Differential plasma profile | Baseline and immediately after the intervention
  Inflammatory proteins

IPD SHARING:
Plan to Share IPD: Undecided
Upon request by e-mail to the principal investigator